CLINICAL TRIAL: NCT03703505
Title: A Phase I, Open-label Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion and to Assess the Absolute Bioavailability of AG-348 in Healthy Male Subjects Following Administration of a Single Oral Dose of [14C]AG-348 and Concomitant Single Intravenous Microdose of [13C6]AG-348
Brief Title: A Study to Evaluate the Absorption, Distribution, Metabolism, Excretion and Absolute Bioavailability of AG-348 in Healthy Male Participants Following Administration of a Single Oral Dose of [14C]AG-348 and Concomitant Single Intravenous Microdose of [13C6]AG-348
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG348-C-009
Record Dates: First submitted 2018-05-24; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-348 (Experimental): On Day 1, participants fasting for at least 10 hours the night before will receive oral AG-348 followed by intravenous (IV) [13C6]AG-348, 1 hour post-oral dose.
  Interventions: Drug: AG-348; Drug: [13C6]AG-348

INTERVENTIONS:
Drug: AG-348 — 120 milligrams (mg) oral capsule, single dose, contains 100 microcuries (μCi) of radio labelled [14C]AG-348.
Drug: [13C6]AG-348 — IV microdose of approximately 100 micrograms (mcg), single dose.

SUMMARY:
This study will assess absorption, distribution, metabolism, excretion and absolute bioavailability of AG-348 in healthy male participants. Potential participants will be screened within 29 days prior to dose administration to determine eligibility. Eligible Participants will be admitted into the Clinical Research Unit (CRU) one day prior to administration of AG-348 and will be confined to the CRU until at least Day 8. If participants are not eligible for discharge on Day 8, they may remain in the CRU up to Day 11. Radiolabelled analytes of AG-348 will be administered in a single oral and intravenous (IV) dose on Day 1. Participants will be required to fast pre-dose, remain in a supine position for 1 hour post-dose and avoid water for 2 hours post-dose.

ELIGIBILITY:
Inclusion Criteria

* Willing and able to provide voluntary written informed consent;
* Males of any race between 18 and 55 years of age, inclusive;
* Body mass index between 18.5 and 29.0 kilograms per meter squared (kg/m2), inclusive, and a total body weight between 50 and 100 kilograms (kg), inclusive;
* In good health;
* Participants will be surgically sterile for at least 90 days or, when sexually active with female partners of childbearing potential, will be required to use a male condom with spermicide from Check-in until 90 days after study drug administration. Sexual intercourse with female partners who are pregnant or breastfeeding should be avoided unless condoms are used from the time of study drug administration until 90 days after study drug administration. Male participants are required to refrain from donation of sperm from Check-in until 90 days after the last dose of study drug;
* Participants who practice true abstinence, because of the participant's lifestyle choice (ie, the participant should not become abstinent just for the purpose of study participation), are exempt from contraceptive requirements. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception. If a participant who is abstinent at the time of signing the informed consent form (ICF) becomes sexually active they must agree to use contraception as described previously;
* Participants who are exclusively in same-sex relationships, contraceptive requirements do not apply. If a participant who is in a same-sex relationship at the time of signing the ICF becomes engaged in a heterosexual relationship, they must agree to use contraception as described previously;
* Willing and able to communicate verbally and in writing with the Investigator and to participate in all scheduled study procedures (including Follow-up procedures) and abide by the study restrictions;
* Agrees to abstain from any alcohol consumption, starting 48 hours before Check-in and continuing until Discharge;
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria

* History of a medical or surgical condition that, in the opinion of the Investigator, may potentially interfere with study drug absorption, distribution, metabolism, and/or excretion (eg, participant has undergone gastrectomy, appendectomy, or cholecystectomy);
* Undergone any major surgical procedure within the past 3 months;
* After 5 minutes of rest in the supine position at Screening, has a systolic blood pressure (BP) reading of ≥140 mmHg (≥150 mmHg in participants >45 years of age) OR a diastolic BP reading of ≥90 mmHg;
* Experienced any serious adverse reaction or serious hypersensitivity to any drug or its formulation excipients;
* History of a primary malignancy, with the exception of a malignancy that has been curatively treated and for which the participant has displayed no evidence of disease within the past 3 years;
* History of alcoholism or drug/chemical abuse within the past 2 years;
* Alcohol consumption of >21 units per week. One unit of alcohol equals 12 oz (360 mL) of beer, 1½ oz (45 mL) of liquor, or 5 oz (150 mL) of wine;
* Positive urine drug screen at Screening or Check-in, or positive alcohol breath test at Check-in (confirmed by repeat);
* Positive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus;
* Participation in a clinical study involving administration of an investigational product (IP) or new chemical entity (NCE) in the past 90 days, or 5 half-lives, if known, of the respective IP or NCE, whichever is longer;
* Has taken, within the 14 days prior to Check-in, any of the following: prescription medication, over-the-counter medication, nonprescription preparation (including vitamins, minerals, phytotherapeutic/herbal/plant-derived preparations), or grapefruit products;
* Has taken within the 28 days prior to Check-in, any restricted product known to strongly induce cytochrome P450 (CYP) 3A4 metabolism (eg, St. John's wort);
* Is a current smoker or user of any other tobacco product, as confirmed by Screening and Check-in urine cotinine test OR has used any tobacco product within the past 3 months
* Receipt of blood products within the past 2 months;
* Donation of blood within the past 56 days, plasma within the past 2 weeks or platelets within the past 6 weeks;
* Previously completed or withdrawn from this study or any other study investigating AG-348, and have previously received the IP;
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures (eg, computed tomography scan, barium meal) exceeding 5 millisieverts (mSv) in the last 12 months or 10 mSv in the last 5 years, or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in;
* Participants who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study.
* Is an employee of, or an immediate family member of an employee of, the study site or the Sponsor;
* Participants who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
AG-348 Excreted Through Urine [A(eu)] | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
AG-348 Excreted through Feces [A(ef)] | Pre-oral dose and 0-24 hr, 24-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Total Amount Excreted Through Urine [Cumulative A(eu)] of AG-348 | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Total Amount Excreted Through Feces [Cumulative A(ef)] of AG-348 | Pre-oral dose and 0-24 hr, 24-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Percentage Excreted in Urine [f(eu)] of AG-348 | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Percentage Excreted in Feces [f(ef)] of AG-348 | Pre-oral dose and 0-24 hr, 24-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Renal Clearance [CL(R)] for AG-348 | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Percentage of Total Radioactivity in Total Excreta (Urine and Feces) | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Area Under the Concentration-Time Curve From Time Zero to the Last Non-Zero Concentration [AUC(0- t)] | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Area Under the Concentration-Time Curve From Time Zero to Infinity Concentration [AUC(0-inf)] | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Maximum Observed Concentration (Cmax) | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Time of Observed Cmax (Tmax) | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Apparent Terminal Elimination Half-life [t(1/2)] | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Ratio of [AUC(0-inf)] of Plasma AG-348 Relative to [AUC(0-inf)] of Plasma Total Radioactivity, [AUC(0-inf)] Plasma AG-348/Total Radioactivity Ratio | Pre-dose and 15, 30, 45, 61, and 90 min and 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, and 144, and 168 hr post-dose
Ratio of [AUC(0-inf)] of Whole Blood Total Radioactivity Relative to [AUC(0-inf)] of Plasma Total Radioactivity, [AUC(0-inf)] Blood/Plasma Ratio | Pre-dose and 15, 30, 45, 61, and 90 min and 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, and 144, and 168 hr post-dose
Total Clearance (CL) of [13C6]AG-348 | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Volume of Distribution [V(z)] of [13C6]AG-348 | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Volume of Distribution at Steady State [V(ss)] for [13C6]AG-348 | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Absolute Bioavailability (F) for AG-348 | Pre-oral dose and 15 min, 30 min, 45 min, 60 min, 61 min, 62 min, 75 min, 90, min 105 min, 2 hr, 3hr, 4 hr, 6 hr, 8 hr, 10 hr, 12, hr 16, hr 24 hr, 36 hr, 48 hr and 72 hr post-oral dose
Plasma Concentrations of AG-348 Metabolites | Pre-dose and 30 min, 61 min, 2 hr, 4 hr, 8 hr, 12 hr, 24, hr, 48 hr, 72 hr, 120 hr and 168 hr post-oral dose

SECONDARY OUTCOMES:
Concentration of AG-348 Metabolites in Urine | Pre-oral dose and 0-4 hours (hr), 4-8 hr, 8-12 hr, 12-24 hr, 24-36 hr, 36-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Concentration of AG-348 Metabolites in Feces | Pre-oral dose and 0-24 hr, 24-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, 120-144 hr and 168 hr post-oral dose
Percentage of Participants Experiencing an Adverse Event | Screening to the end of study (up to 40 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Covance, Madison, Wisconsin, United States